CLINICAL TRIAL: NCT04789642
Title: Effect of an Educational Program Using Virtual Social Network on Nurses' Knowledge and Skill of Blood Pressure Measurement
Brief Title: Nurses Education Using Virtual Social Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, mohamed elsayed hamed elzeky, lecturer, medical surgical nursing department, faculty of nursing, Mansoura university, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: mansoura U
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Blood Pressure Determination; Continuing Nursing Education; Education, Distance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): A social group will be created on whatsapp for subjects of the intervention group and they will receive education about blood pressure measurement guidelines in 24 sessions, once per day in the form of text, image and video clips. In addition to British and Irish Hypertension Society (BIHS) blood pressure measurement auscultatory tutorials.
  Interventions: Other: blood pressure measurement whatsapp educational program
- control group (No Intervention): The control group will not receive any intervention only their routine education that is provided by the continuous staff development team of the hospital.

INTERVENTIONS:
Other: blood pressure measurement whatsapp educational program — educational
  Arms: study group

SUMMARY:
Regardless of the method used to measure BP, initial and ongoing training of technicians and healthcare providers and the use of validated and calibrated devices are critical for obtaining accurate BP measurements.

DETAILED DESCRIPTION:
Shortage of human resources and the importance of remaining up-to-date to provide healthcare services highlighted the development of distance education for nurses. In addition information presented via the distance learning method via software systems was more stable than the face-to-face method via lecture, and it saved time and energy. Nurses are responsible for BP monitoring and assessment in the clinical setting. Finding new strategies for distance education is of great concern and ,compared with traditional face-to-face interventions, those carried out through social networks have the advantage that the participant does not need to attend the sessions in person, and offers unlimited access to the intervention materials whenever they wish.

ELIGIBILITY:
Inclusion Criteria:

* Only permanent staff nurses working in the two cardiac units.
* Nurses of both sexes .
* Nurses who use a smart phone or any other digital device with the ability to install the social network of whatsapp.

Exclusion Criteria:

* Inaccessibility to wireless net work
* Unwillingness to participate in study
* Failure to fill pretest questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
change in blood pressure measurement skill score | will be measured at baseline and at the end of study (after 1 month)
  ). It consists of nine parts. Part one focuses on participants' ability to correctly identify the Korotkoff soundsParts two to nine will focus on measurement steps and a scoring system will be applied by adding 1 point to each correct practice, and 0 point to each wrong practice
change in Blood Pressure Measurement Knowledge score | will be measured at baseline and at the end of the study (after 1 month)
  It consists of five sections. Section one focuses on demographic information , Section two to five focus on questions related to background knowledge, measurement technique, cuff size and arm position of the patient, palpation to identify systolic pressure. A scoring system will be applied by adding 1 point to each correct answer, and 0 point to each wrong answer.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elzeky MEH, Shahine NFM. Effects of an educational program using a virtual social network on nurses' knowledge and performance of blood pressure measurement: a randomized controlled trial. BMC Nurs. 2022 Dec 21;21(1):365. doi: 10.1186/s12912-022-01137-0. PMID 36544166